CLINICAL TRIAL: NCT04779047
Title: Comparative Therapeutic Efficacy and Safety of Remdesivir Plus Lopinavir/ Ritonavir and Tocilizumab Versus Hydroxychloroquine Plus Ivermectin and Tocilizumab in COVID-19 Patients.
Brief Title: Comparative Therapeutic Efficacy and Safety of Different Antiviral and Anti Inflammatory Drugs in COVID-19 Patients.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: October 6 University (Other)
Collaborators: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Ahmed Essam, Principle Investigator, October 6 University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC-H-PhBSU-21011
Record Dates: First submitted 2021-02-25; First posted 2021-03-03 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Covid19; Pneumonia
Keywords: covid19
MeSH Terms: conditions — COVID-19; Pneumonia | interventions — remdesivir; Hydroxychloroquine; tocilizumab; Lopinavir; lopinavir-ritonavir drug combination; Ivermectin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- group 1 (Active Comparator): Remdesivir will be administrated intravenously (IV) at a dose of 200 mg at day 1 then 100 mg once daily for 5 days and Lopinavir / ritonavir at a dose of 400 /100 once daily for 5 days plus tocilizumab 800 mg once
  Interventions: Drug: Remdesivir; Drug: Tocilizumab; Drug: Lopinavir/ Ritonavir
- group 2 (Active Comparator): Hydroxychloroquine will be administrated at a dose of 400 mg twice daily at day 1 then 200 mg twice daily for 5 days and Ivermectin 36 mg at day 1,3 and 6 plus tocilizumab 800 mg once.
  Interventions: Drug: Hydroxychloroquine; Drug: Tocilizumab; Drug: Ivermectin

INTERVENTIONS:
Drug: Remdesivir — Remdesivir will be administrated intravenously (IV) at a dose of 200 mg at day 1 then 100 mg once daily for 5 days.
  Arms: group 1
Drug: Hydroxychloroquine — Hydroxychloroquine will be administrated at a dose of 400 mg twice daily at day 1 then 200 mg twice daily for 5 days.
  Arms: group 2
Drug: Tocilizumab — Tocilizumab 800 mg once.
  Other Names: Actemra
Drug: Lopinavir/ Ritonavir — Lopinavir / ritonavir at a dose of 400 /100 once daily for 5 days.
  Other Names: kaletra
  Arms: group 1
Drug: Ivermectin — Ivermectin 36 mg at day 1,3 and 6.
  Other Names: Iverazine
  Arms: group 2

SUMMARY:
Comparison outcomes of a large cohort of moderate and severe COVID-19 patients received different Antiviral and Anti Inflammatory Drugs.

DETAILED DESCRIPTION:
Aim of the study

1. To assess the difference in patients' clinical status improvement between patients.
2. To detect time to improvement in oxygenation among both groups.
3. To detect duration of hospitalization and mortality rate in both groups.
4. To detect incidence and duration of mechanical ventilation in both treatment arms.
5. To monitor of adverse events of both drugs

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized adult patients with pneumonia evidenced by chest CT scan.
* Laboratory (RT-PCR) confirmed infection with 2019-nCoV or strongly suspected to be infected with SARS-COV2 with confirmation studies pending.
* And at least one of the following:

  1. Respiratory frequency ≥30/min.
  2. Blood oxygen saturation ≤93% on room air (RA).
  3. Partial pressure of arterial oxygen to fraction of inspired oxygen ratio (PaO2/FiO2) <300.
  4. Worsening of lung involvement, defined as an increase in number and/or extension of pulmonary areas of consolidation, need for increased FiO2 to maintain stable O2 saturation, or worsening O2 saturation of >3% with stable FiO2.

Exclusion Criteria:

* Baseline elevation of alanine aminotransferase (ALT) or aspartate aminotransferase (AST) levels > 3-fold the upper limit of the normal range.
* Pregnancy.

Ages: 18 Years to 88 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-03-10 (Estimated); Study Completion 2021-04-05 (Estimated)

PRIMARY OUTCOMES:
Percentage of clinical cure in each arm | through an average of 5-7 days
  Proportion of cured patients in the interventional group versus the proportion of cured patients in the control group before and after starting drugs

CONTACTS AND LOCATIONS:
Overall Officials: Marian Boshra, PhD, Principal Investigator — Beni-Suef University
Locations (1):
- Beni-suef University, Banī Suwayf, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sarhan RM, Harb HS, Abou Warda AE, Salem-Bekhit MM, Shakeel F, Alzahrani SA, Madney YM, Boshra MS. Efficacy of the early treatment with tocilizumab-hydroxychloroquine and tocilizumab-remdesivir in severe COVID-19 Patients. J Infect Public Health. 2022 Jan;15(1):116-122. doi: 10.1016/j.jiph.2021.10.024. Epub 2021 Nov 2. PMID 34764044